CLINICAL TRIAL: NCT03792295
Title: The Effect of Multimodal Pain Therapy After Hernia Repair
Brief Title: Multimodal Pain Therapy After Hernia Repair
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no enrollment, reallocation of resources
Sponsor: Khashayar Vaziri (Other)
Responsible Party: Sponsor-Investigator, Khashayar Vaziri, Associate Professor of Surgery, George Washington University
Organization: George Washington University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MultimodalHernia
Record Dates: First submitted 2018-12-27; First posted 2019-01-03 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Hernia, Abdominal; Pain
MeSH Terms: conditions — Hernia, Abdominal; Pain | interventions — Acetaminophen; Ibuprofen; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multimodal Therapy (Experimental): Patients will receive scheduled ibuprofen 400mg po q 4 hours and acetominophen 1gram po q 8 hours during the post operative phase and oxycodone 5mg po q 4 to 6 hours as needed for pain control.
  Interventions: Drug: acetominophen, ibuprofen, oxycodone
- Classic/standard opiod Therapy (Active Comparator): Patients will receive oxycodone 5mg po q 4 to 6 hours as needed during their post operative phase for pain control.
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: acetominophen, ibuprofen, oxycodone — Multimodal pain treatment group
  Other Names: Tylenol, Advil, OxyContin
  Arms: Multimodal Therapy
Drug: Oxycodone — Classic opiod pain treatment group
  Other Names: OxyContin
  Arms: Classic/standard opiod Therapy

SUMMARY:
Investigating the effect of multimodal pain treatment after hernia repair

DETAILED DESCRIPTION:
This is a randomized, non-blinded study comparing the effects of multimodal pain management (ibuprofen, tylenol, and narcotics/oxycodone as needed) for relief of post-operative pain in patients who undergo hernia repair. Patients who present for elective hernia surgery will be randomized in a 1:1 fashion by pre-operative pain score into a multimodal pain treatment group or conventional opiod treatment group for post-operative pain management. They will be followed up after their surgery to evaluate their pain scores and narcotic use.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult patients >18 years of age to 90 years of age who are eligible for a hernia repair (ventral or inguinal) by a surgeon in the Medical Faculty Associates Department of General Surgery at the George Washington University Hospital.

Exclusion Criteria:

* Patients with allergies to sulfa or any of the medications being evaluated in this study (ibuprofen, tylenol, oxycodone)
* patients with a history of gastric ulcer or gastrointestinal bleeding
* patients with kidney disease
* patients with cardiovascular disease
* patients with a co-morbid condition that would prohibit them from taking narcotics
* patients with known or suspected narcotic abuse
* patients who do not wish to participate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Post operative pain scores at rest and during movement | 1-14 days after surgery
  Patients will be called on post operative days 1-3 and asked to rate their pain while at rest and during movement using the following scales:
  On a scale of 1-10, with 1=no pain and 10= the worst pain, what has been your average pain level since surgery during REST? 1 2 3 4 5 6 7 8 9 10
  On a scale of 1-10, with 1=no pain and 10= the worst pain, what has been your average pain level since surgery during MOVEMENT (such as walking across the room)? 1 2 3 4 5 6 7 8 9 10
  Patients will also be asked the same two pain scales (pain at rest and during movement) at the first post-operative appointment, which will occur within 14 days of their surgery.
  The scores for pain at rest and during movement will not be summed or averaged together, so that the maximum score on each scale is 10 (worst pain), and the minimum score is 1 (no pain). Scores will not be summed across days. Lower scores are considered a better outcome, and higher scores are considered a worse outcome.

SECONDARY OUTCOMES:
Narcotic use | 1-14 days after surgery
  Amount of oxycodone pills taken

CONTACTS AND LOCATIONS:
Locations (1):
- George Washington University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rudd RA, Seth P, David F, Scholl L. Increases in Drug and Opioid-Involved Overdose Deaths - United States, 2010-2015. MMWR Morb Mortal Wkly Rep. 2016 Dec 30;65(50-51):1445-1452. doi: 10.15585/mmwr.mm655051e1. PMID 28033313
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Manworren RC. Multimodal pain management and the future of a personalized medicine approach to pain. AORN J. 2015 Mar;101(3):308-14; quiz 315-8. doi: 10.1016/j.aorn.2014.12.009. PMID 25707723
- [Background] Warren JA, Stoddard C, Hunter AL, Horton AJ, Atwood C, Ewing JA, Pusker S, Cancellaro VA, Walker KB, Cobb WS, Carbonell AM, Morgan RR. Effect of Multimodal Analgesia on Opioid Use After Open Ventral Hernia Repair. J Gastrointest Surg. 2017 Oct;21(10):1692-1699. doi: 10.1007/s11605-017-3529-4. Epub 2017 Aug 14. PMID 28808868
- [Background] Majumder A, Fayezizadeh M, Neupane R, Elliott HL, Novitsky YW. Benefits of Multimodal Enhanced Recovery Pathway in Patients Undergoing Open Ventral Hernia Repair. J Am Coll Surg. 2016 Jun;222(6):1106-15. doi: 10.1016/j.jamcollsurg.2016.02.015. Epub 2016 Mar 3. PMID 27049780
- [Background] Fayezizadeh M, Petro CC, Rosen MJ, Novitsky YW. Enhanced recovery after surgery pathway for abdominal wall reconstruction: pilot study and preliminary outcomes. Plast Reconstr Surg. 2014 Oct;134(4 Suppl 2):151S-159S. doi: 10.1097/PRS.0000000000000674. PMID 25254998